CLINICAL TRIAL: NCT04255082
Title: Mindfulness and Shared Decision Making
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 030.HEP.2018.D
Record Dates: First submitted 2019-04-03; First posted 2020-02-05 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assess the impact of mindfulness-based interventions on inpatients' and outpatients' stress, patient-provider communication, and other measures of SDM at MDMC. — Effectiveness of the mindfulness-based intervention which will be assessed by:
  Baseline and post-intervention perception of stress and anxiety Impact of stress on communication Emotional/Brain state Level of SDM during a pivotal visit with provider e.g. treatment planning visit (for outpatients only) The Emotional Distress-Anxiety (PROMIS, 2016), Communication Short Form (Cella, PROMIS, 2013), Emotional/Brain State Question (Mellin, 2017) and The Shared Decision Making dyadic OPTION scale (Melbourne, 2016) will be used to evaluate these outcomes.
  Feasibility of such a study in the patient population and setting. This will be measured by the barriers encountered and the ability to successfully carry out the study.

SUMMARY:
The purpose of this study is to assess the impact of mindfulness-based interventions on patient stress, patient-provider communication, and other measures of SDM at MDMC.

There is a need to have a quantifiable measure of perceived stress and communication ability in patients. This is the first study of its kind to be conducted at MDMC. This pilot study will not only benefit the patients but also contribute to the medical community's understanding of treating the whole patient through mindfulness and shared decision making.

2.1. Study Objectives 2.1.1. Primary Objective To assess the impact of mindfulness-based interventions on inpatients and outpatients stress, patient-provider communication, and other measures of SDM at MDMC.

2.1.2. Secondary Objectives To evaluate the feasibility of such a study in the patient population.

DETAILED DESCRIPTION:
This will be a prospective cohort of patients at MDMC, The Liver Institute, and Texas Oncology between 6/1/2018 and 12/31/2020. Subject records will be reviewed to identify case-based details including demographics, diagnosis, and date of diagnosis. Subjects will complete survey instruments to assess their levels of stress and anxiety, and the impact of the same on their ability to communicate at baseline, after the stress management coaching session, following their treatment planning visit (outpatients only), and one week after the visit (by mail). Providers will also complete the dyadic OPTION instrument (for outpatients only) to empirically assess the perceived degree of patient involvement in the treatment planning process. The face-to-face stress management coaching session will occur approximately an hour before meeting with the treatment planning team for outpatients and at a designated time identified for inpatients. The session will focus on mindfulness-based interventions on stress regulation, communication, and shared decision making. A comprehensive evaluation will be performed and a unique treatment plan developed for each subject based on a biopsychosocial model to address the mind, body, and spirit. Nutritional counseling and lifestyle coaching will also be addressed.

2.2. Study Outcome Measures 2.2.1. Primary Outcome

The effectiveness of the mindfulness-based intervention which will be assessed by:

Baseline and post-intervention perception of stress and anxiety Impact of stress on communication Emotional-Brain state Level of SDM during a pivotal visit with provider e.g. treatment planning visit (for outpatients only) The Emotional Distress-Anxiety (PROMIS, 2016), Communication Short Form (Cella, PROMIS, 2013), Emotional/Brain State Question (Mellin, 2017) and The Shared Decision Making dyadic OPTION scale (Melbourne, 2016) will be used to evaluate these outcomes.

2.2.2. Secondary Outcome Feasibility of such a study in the patient population and setting. This will be measured by the barriers encountered and the ability to successfully carry out the study.

2.3 Study Enrollment: 2.3.1.Study Inclusion Criteria

* Age 18 years or olde
* Newly diagnosed cancer patient (breast, pancreatic, head & neck, hepatocellular carcinoma, cholangiocarcinoma, and colorectal carcinoma with metastases to the liver) at MDMC, the Liver Institute, or Texas Oncology
* Provided written informed consent 2.3.2. Study Exclusion Criteria
* Below 18 years of age
* Does not have cancer

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Inpatients and outpatients receiving treatment at MDMC, the Liver Institute, or Texas Oncology
* Provided written informed consent

Exclusion Criteria:

* Below 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at MDMC, The Liver Institute, and Texas Oncology between 6/1/2018 and 12/31/2020.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Baseline and post-intervention perception of stress & anxiety by answering survey questions | 6/1/2018 and 12/31/2020
  Effectiveness of the mindfulness-based intervention which will be assessed by survey questions:
  Baseline and post-intervention perception of stress and anxiety t of stress on communication Emotional/Brain state Level of SDM during a pivotal visit with provider e.g. treatment planning visit (for outpatients only) The Emotional Distress-Anxiety (PROMIS, 2016).

SECONDARY OUTCOMES:
Feasibility of a study in the patient population and setting by any difficulties faced during the study phase | 6/1/2018 and 12/31/2020
  Feasibility of such a study in the patient population and setting. This will be measured by the barriers encountered and the ability to successfully carry out the study. The study questionnaire will be used for the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, M.D., Principal Investigator — Methodist Health System
Locations (1):
- The Liver Institute at Methodist Dallas Medical Center, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No